CLINICAL TRIAL: NCT04569981
Title: Climb up, Heads up: Sport Climbing With Parkinson's Disease
Brief Title: Sport Climbing With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Vienna (Other); University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Heidemarie Zach, MD, BSc., Principal Inversigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1369/2017
Record Dates: First submitted 2020-08-17; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; sport climbing; motor symptoms; training therapy
MeSH Terms: conditions — Parkinson Disease | interventions — Stair Climbing

STUDY DESIGN:
Intervention Model Description: The participants were randomly assigned to either the climbng group or the unsupervised active group
Who Masked: Care Provider
Masking Description: Movement disorder specialists who performed the MDS-UPDRS III ratings were blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Climbing Group (CG) (Active Comparator): The patients in the Climbing Group (CG) followed a 12-weeks long climbing trainings course in small groups of 3-4 participants with a certified climbing instructor.
  Interventions: Other: Climbing
- Unsupervised active group (UAG) (Active Comparator): The patients in the unsupervised activity group (UAG) received education European physiotherapy guidelines for physical activity recommended by the WHO of recommended activity and followed their self-selected activities over 12 weeks.
  Interventions: Other: Unsupervised activity group

INTERVENTIONS:
Other: Climbing — The patients in the Climbing Group (CG) followed a 12-weeks long climbing trainings course in small groups of 3-4 participants with a certified climbing instructor.
  Arms: Climbing Group (CG)
Other: Unsupervised activity group — The patients in the unsupervised activity group (UAG) received education European physiotherapy guidelines for physical activity recommended by the WHO of recommended activity and followed their self-selected activities over 12 weeks.
  Arms: Unsupervised active group (UAG)

SUMMARY:
This controlled interventional study will investigate the effects of a 12-weeks sport climbing course compared to 24 weeks of unsupervised physical exercise on motor symptoms in Parkinson's disease

DETAILED DESCRIPTION:
The primary aim of this study is to evaluate the effects of a 12-week sport climbing course versus unsupervised physical exercise on motor symptoms in patients with Parkinson's disease.

Background: Sport climbing (SC) is known as a whole-body workout, which additionally trains cognitive, mental, and social abilities. In contrast to its public image, SC in a controlled environment using "top-rope" belay, is a safe sport and can be performed at any age and at any level. In the field of neurological rehabilitation, it is already used as "therapeutic SC" for other neurological diseases, such as stroke, multiple sclerosis, depressions etc. but studies on climbing in PD patients are lacking.

Hypothesis: to find significant improvement of motor symptoms in the climbing group compared to the control group as well as biopsychosocial improvements after 6 weeks, 12 weeks, and 6 months after the intervention.

Methods: Effects of SC on motor symptoms in 48 PD patients in total, who will be randomized into a climbing group (n=24) and a control group (n=24) will be evaluated. The climbing group will follow a 12-week 90 min/week climbing trainings course, led by professional climbing instructors.

The control group will receive education/information material of the European physiotherapy guidelines for physical activity recommended by the WHO and will be instructed to follow the recommendation of the guidelines to independently live an active lifestyle and train unsupervised. All patients will be evaluated with clinical assessments at baseline, in between the study period (mid), after completing the 12-weeks study period (post). As additional outcomes, health benefits of SC in PD with a holistic approach, covering biopsychosocial aspects will be investigated. Therefore, non-motoric and motoric parameters will be evaluated, and follow-up assessments 6 months after.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* HY stage 1-3

Exclusion Criteria:

* cognitive impairment
* severe hearing or visual impairment
* severe orthopedic problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
Clinical Rating | Testpoints: Change from Baseline Score after 12 weeks of the intervention
  Motor Part of the Movement Disorders Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) III

SECONDARY OUTCOMES:
Change in Gait and Balance using wearable sensors | Testpoints: Change after 12 weeks of the intervention
  Inertial Sensors will be used to quantify gait metrics (postural sway, gait cycle, speed) as participants conduct walking and balance trials
Quantified Bradykinesia test | Testpoints: Change after 12 weeks of the intervention
  Changes in a quantified bradykinesia Tests by using a standardized speeded keyboard tapping task. Changes will be evaluates in keys/second
Hand grip strength | Testpoints: Change after 12 weeks of the intervention
  Assessment of hand grip strength, using a dynamometer. Results will be evaluated in Kilogramms
Parkinson Quality of Life Questionaire-39 (PDQ-39) | Testpoints: Change after 12 weeks of the intervention
  Quality of life, assessed by the PDQ-39 Questionnaire
Social Outcomes | Testpoints: Change after 12 weeks of the intervention
  Questionnaiers about social effects
Cognitive assessments | Testpoints: Change after 12 weeks of the intervention
  Change in cognition will be assessed using a standardized cognitive assessment battery, measuring following domains: executive functions, memory, attention and verbal functions
Changes in brain functional and structural MRI (resting state paradigma) and Changes in brain structural and functional MRI | Testpoints: Change after 12 weeks of the intervention
  Changes in structural and functional MRI (resting state paradigma) will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Neurology, Vienna, Austria

REFERENCES:
- [Derived] Langer A, Hansen C, Roth D, Santer A, Flotz A, Gruber J, Wizany L, Hasenauer S, Pokan R, Dabnichki P, Treven M, Zimmel S, Schmoeger M, Willinger U, Gassner L, Brucke C, Maetzler W, Zach H. Vertical locomotion improves horizontal locomotion: effects of climbing on gait and other mobility aspects in Parkinson's disease. A secondary analysis from a randomized controlled trial. J Neuroeng Rehabil. 2024 Apr 27;21(1):63. doi: 10.1186/s12984-024-01363-4. PMID 38678241